CLINICAL TRIAL: NCT02929173
Title: Patient Satisfaction and Clinical Assessment of Biocompatible High Performance Polymers Crown Veneered With Visio.Lign Versus E-max Crown Veneered With E-max Veneering System in Anterior Aesthetic Zone.(Randomized Controlled Clinical Trial)
Brief Title: Effect of Different Types of Crowns on Patient Satisfaction and Clinical Assesment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora helmy hassaneen, assistant lecturer of fixed prosthodontic department,MTI university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-217
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Personal Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — AllCeram

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Active Comparator): E-max is un allceram crown
  Interventions: Other: Allceram
- Group 1 (Experimental): Bio HPP crown is a hybrid crown
  Interventions: Other: hybrid crown

INTERVENTIONS:
Other: Allceram — Pressed E-max coping veneered with E-max veneering system
  Other Names: Prosthetic Crown
  Arms: Group 2
Other: hybrid crown — pressed Bio HPP coping veneered with visolign veneering system
  Other Names: Prosthetic Crown
  Arms: Group 1

SUMMARY:
The aim of this study is to compare the patient satisfaction and clinical assessment (shade matching, surface texture and marginal discoloration) of Bio- High Performance Polymers (HPP) restoration versus E-max restoration compared to contralateral tooth in anterior zone.

Regardless E-max popularity in the dental field.

DETAILED DESCRIPTION:
Roles and responsibilities

1. Nora Helmy Hasaneen (N.H.): Operator, data enterer and corresponding author; Assistant lecturer fixed Prosthodontics Department, Faculty of Dentistry, Modern Technology Institution (MTI) University, Egypt.
2. Dr. Ahmed Naguib Hussin( A.H.): Main supervisor, data monitoring and auditing; Professor of fixed Prosthodontics, Faculty of Oral and Dental Medicine- Cairo University, Egypt.
3. Dr.Gihan Al-Naggar (A. G.):Co-Supervisor, data monitoring and auditing; Professor of fixed Prosthodontics, Faculty of Oral and Dental Medicine -Cairo University, Egypt.

3.Esraa Mohamed Odeuh(E.O.):Outcome assessors and data collection; Assistant lecturer, Fixed Prosthodontics Department, Faculty of Oral and Dental Medicine, MTI University, Egypt.

4.Ahmed Gamal(A.G): Base line data collection, recruitment, sequence generation, allocation concealment, patient retention and taking participants' consents; Resident Fixed Prosthodontics Department, Faculty of Oral and Dental Medicine, MTI University, Egypt.

5.Eman Desouky (E.D.):Sample size calculation; Statistician, Faculty of Oral and Dental Medicine, Cairo University, Egypt.

6. Evidence Based Dentistry Committee (CEBD) Help in reporting study protocol following SPIRIT guidelines; Faculty of Oral and Dental Medicine, Cairo University, Egypt.

7.Research Ethics Committee (CREC): Protocol reviewer of the clinical trial in order to protect the right, safety, dignity and well-being of the participants; Faculty of Oral and Dental Medicine, Cairo University, Egypt.

8. Research Plan Committee (CRPC):For ensuring that this clinical trial following the department research plan; Fixed prosthodontic Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.

1. Intervention:

   N.H. will perform conservative tooth preparation following the principles of all ceramic crown preparation with shoulder subgingival finish line of thickness 1.2mm using tapered stone with flat end attached to high speed headpiece with air and water coolant, after local anesthesia has been given.

   N.H. will take adequate 2ry Impression using non aqueous Elastomeric impression materials Impregum™F (medium consistency, 3M ESPE ,) and bite registration will by pink soft wax (Stardentalsupply) .

   N.A. & E.O. will visually select the shade match using Vita Easyshade Compact (Vita Zahnfabrik, Bad Sa¨ckingen,Germany). N.H will fabricate the temporary restoration using Protemp™ 4 Temporisation Material(3M ESPE ) and cemented using non Eugenol Zinc Oxide temporary cement TempBond™ Temporization (Kerrdentalsupply).

   N.H will deliver Press Bio - HPP framework material veneered with visio lign veneering material (Bredent) crown and cement it with 3M™ ESPE™ RelyX™ Unicem Self-Adhesive Universal Resin Cement.
2. Comparator N.H. will perform conservative tooth preparation following the principles of all ceramic crown preparation with shoulder subgingival finish line of thickness 1.2mm using tapered stone with flat end attached to high speed headpiece with air and water coolant, after local anesthesia has been given.

   N.H. will take adequate 2ry Impression using non aqueous Elastomeric impression materials Impregum™F (medium consistency, 3M ESPE ,) and bite registration will by pink soft wax (Stardentalsupply) .

   N.A. & E.O. will visually select the shade match using Vita Easyshade Compact (Vita Zahnfabrik, Bad Sa¨ckingen,Germany). N.H will fabricate the temporary restoration using Protemp™ 4 Temporisation Material(3M ESPE ) and cemented using non Eugenol Zinc Oxide temporary cement TempBond™ Temporization (Kerrdentalsupply).

   N.H will deliver E.max® framework veneered with E-max veneering System (Ivoclar Vivadent) crown and cement it with 3M™ ESPE™ RelyX™ Unicem Self-Adhesive Universal Resin Cement.
3. Outcomes

A. Primary outcome: Patient satisfaction:

E.O will measure patient satisfaction using Rating scores. The mean and standard deviation for the Rating scores of the patients will be recorded at the time of crown cementation, 3, 6, 9 & 12 months after review for aesthetics.

B. Secondary outcome: Clinical assessment of the restoration:

E.O will evaluate shade matching, marginal discoloration and surface texture using modified USPHS criteria scores. The mean and standard deviation for the USPHS criteria scores of the patients will be recorded at the time of crown cementation 0, 3, 6, 9 & 12 months after review for aesthetics.

ELIGIBILITY:
Inclusion Criteria:

1. Patient will be able to physically and psychologically to tolerate conventional restorative procedures.
2. Patients have no active periodontal or pulpal diseases, have teeth with good restorations.
3. Patient with anterior tooth with problems indicated for full coverage restoration (e.g. mild to moderate discoloration, coronal fracture where partial coverage would lack retention, malposed or malformed teeth) Patients are willing to return for follow-up examination and evaluation.
4. Patient with sound contralateral tooth to the selected tooth required for full coverage.
5. Patient with root canal treated tooth requiring full coverage restoration

Exclusion Criteria:

1. Patient in the growth stage with partially erupted teeth.
2. Patient with poor oral hygiene and motivation.
3. Pregnant women's.
4. Patient with psychiatric problems or unrealistic expectations.
5. Patients have no opposing occluding dentition in the area intended for restoration.
6. Patients with parafunctional habits.
7. Color blindness patients are excluded.
8. Patient without contralateral tooth to that tooth to will be restored.
9. Patient without adjacent teeth to that tooth will be restored.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in esthetic patient satisfaction | At crown delivery time and after delivery 3, 6, 9, 12 month
  using Rating scores from 0-2 (0= Poor, 1=Accepted, 2=Excellent)

SECONDARY OUTCOMES:
Shade match to contralateral tooth | At crown delivery time and after delivery 3, 6, 9, 12 month
  using Modified USPHS scores from 0-3 (0= Match to contralateral tooth, 1=Acceptable mismatch to contralateral tooth , 2=Unacceptable mismatch to contralateral tooth, 3=New restoration is needed.)
Marginal discolouration | At crown delivery time and after delivery 3, 6, 9, 12 month
  using Modified USPHS scores from 0-3 (0= Smooth surface., 1=Slight staining can be polished away., 2=Gross staining., 3=New restoration is needed.)
Surface texture | At crown delivery time and after delivery 3, 6, 9, 12 month
  using Modified USPHS scores from 0-3 (0= Surface is smooth as the surrounding., 1=Surface is rough than the surrounding, 2=Gross staining., 3=Surface is very rough avoiding movement of the explorer, 4=New restoration is needed.)

IPD SHARING:
Plan to Share IPD: No